CLINICAL TRIAL: NCT02838810
Title: The Optimizing Treatment of PegIFN Alfa in HBeAg-negative Chronic Hepatitis B Patients With Low Level HBsAg
Brief Title: The Optimizing Treatment of PegIFN Alfa in HBeAg-negative CHB Patients With Low Level HBsAg
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Peking University (Other); Shenzhen Third People's Hospital (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, Chief director of department of infectious disease, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-Cure-2
Record Dates: First submitted 2016-07-16; First posted 2016-07-20 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis B
Keywords: peginterferon alfa; Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — nas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): CHB patients with low level HBsAg.Hepatitis B e antigen (HBeAg)-negative CHB patients who had received NAs for more than 12 months, with HBsAg <1000 IU/mL and Hepatitis B virus DNA <100 IU/mL, are to receive peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week. The longest course of treatment is 96 weeks. After treatment, patients will be followed up for 24 weeks. During the 96 weeks course of treatment, HBsAg level will be monitored. When HBsAg level is less than 0.05 IU/mL, peginterferon treatment will be stopped and patients will receive 24 weeks follow up.
  Interventions: Drug: peginterferon alfa
- Control (Other): Patients do not need to change their NAs treatment.
  Interventions: Drug: Nucleoside analogues

INTERVENTIONS:
Drug: peginterferon alfa — peginterferon alfa-2b or peginterferon alfa-2a
  Arms: Experimental
Drug: Nucleoside analogues — Nucleoside analogues
  Other Names: NAs
  Arms: Control

SUMMARY:
As HBsAg clearance is uncommon in chronic hepatitis B (CHB) patients on nucleoside analogues (NAs) therapy. The purpose of this study is to optimize HBsAg clearance in CHB Patients with sequential treatment of pegylated interferon alpha and NAs.

DETAILED DESCRIPTION:
In order to optimize HBsAg clearance in CHB patients with low level HBsAg, the investigators enrolled patients who had received, and responded to, NAs for more than 12 months(see the inclusion criteria), and patients are switched to receive peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week. The longest course of treatment is 96 weeks. After treatment, patients will be followed up for 24 weeks. During the 96 weeks course of treatment, HBsAg level will be monitored. When HBsAg level is less than 0.05 IU/mL, peginterferon treatment will be stopped and patients will receive 24 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

1. CHB patients who had received single NAs for more than 12 months.
2. Hepatitis B e antigen (HBeAg)-negative.
3. Hepatitis B surface antigen (HBsAg) positive and <1000 IU/mL.
4. Hepatitis B virus DNA <100 IU/mL.

Exclusion Criteria:

1. Patients with liver cirrhosis, Hepatocellular Carcinoma or AFP >2 ULN or other malignancies.
2. Patients with other factors causing liver diseases.
3. Pregnant and lactating women.
4. Patients with concomitant HIV infection or congenital immune deficiency diseases.
5. Patients with diabetes, autoimmune diseases.
6. Patients with important organ dysfunctions.
7. Patients with serious complications (e.g., infection, hepatic encephalopathy, hepatorenal syndrome, gastrointestinal bleeding.)
8. Patients who receive antineoplastic or immunomodulatory therapy in the past 12 months.
9. Patients with a previous use of IFN anti hepatitis B virus treatment or have NAs drug resistance.
10. Patients who can't come back to clinic for follow-up on schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
HBsAg Clearance | 120 weeks
  Percentage of Participants with HBsAg <0.05 IU/mL.
HBsAg Seroconversion | 120 weeks
  Percentage of Participants with HBsAg <0.05 IU/mL and anti-HBsAg positive.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiliang Gao, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The third affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided